CLINICAL TRIAL: NCT01557777
Title: An Extension Study of Navitoclax (ABT-263) in Subjects With Chronic Lymphocytic Leukemia (CLL)
Brief Title: Open-label Extension Study of Navitoclax in Subjects With Chronic Lymphocytic Leukemia (CLL)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AbbVie (prior sponsor, Abbott) (Industry)
Responsible Party: Sponsor
Organization: AbbVie (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: M13-641; 2012-000606-29 (EudraCT Number)
Record Dates: First submitted 2012-03-16; First posted 2012-03-20 (Estimated); Last update posted 2014-07-04 (Estimated); Status verified 2014-07

CONDITIONS: Chronic Lymphocytic Leukemia
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — navitoclax

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Navitoclax, ABT-263 (Experimental)
  Interventions: Drug: Navitoclax

INTERVENTIONS:
Drug: Navitoclax — QD
  Other Names: ABT-263

SUMMARY:
Open-label extension study of navitoclax in subjects with chronic lymphocytic leukemia (CLL).

DETAILED DESCRIPTION:
This is an open-label extension study of navitoclax in subjects with chronic lymphocytic leukemia (CLL).

ELIGIBILITY:
Inclusion Criteria:

* The subject has been dosing in Arm C of the ABT4710n study, has not discontinued for any reason prior to study closure and the investigator believes that continued treatment with navitoclax is in the best interest of the subject
* The subject must meet defined hematology and coagulation lab criteria as specified in the protocol
* The subject must meet defined chemistry criteria as specified in the protocol
* Women of childbearing potential and men must agree to use adequate contraception (as per protocol) prior to study entry, for the duration of study participation and up to 90 days following completion of therapy
* The subject is capable of understanding and complying with parameters as outlined in the protocol and able to sign the Informed Consent Form

Exclusion Criteria:

* The subject discontinued navitoclax administration in Arm C of the ABT4710n study for reasons of disease progression, Adverse Event toxicity, withdrawal of consent or Investigator decision prior to study completion.
* The subject has any medical condition which in the opinion of the investigator places the subject at an unacceptably high risk for toxicities.
* The subject is a lactating or pregnant female.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2012-06; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Safety: Adverse Events - The number of participants with adverse events will be reported as a measure of Safety. | Adverse events occuring through the Final Visit (up to Week 52) will be reported
  The investigators will monitor each subject for clinical and lab evidence of adverse events on a routine basis through out the study. The investigators will question each subject regarding any adverse effects that they have experienced and record any events on the care report forms. All adverse events will be followed to a satisfactory clinical resolution.
Safety: Physical Examination and Vital Signs - Physical examination will be performed and vital signs will be assessed for participants as a measure of safety. | Change from baseline through Final Visit (up to Week 52).
  Physical exam, blood pressure, pulse, body temperature will be measured and recorded
Safety: Clinical Lab Tests will be performed for each participant as a safety measure. | Change from baseline through Final Visit (up to Week 52).
  Chemistry, hematology, urinalysis lab tests will be measured and recorded. All clinically significant values will be followed by the investigator to a satisfactory clinical resolution.

CONTACTS AND LOCATIONS:
Overall Officials: Mack Mabry, MD, Study Director — AbbVie
Locations (15):
- United States (5):
  - Site Reference ID/Investigator# 74036, La Jolla, California
  - Site Reference ID/Investigator# 74035, Los Angeles, California
  - Site Reference ID/Investigator# 74038, Pleasant Hill, California
  - Site Reference ID/Investigator# 74039, Santa Maria, California
  - Site Reference ID/Investigator# 74033, Bethesda, Maryland
- Australia (2):
  - Site Reference ID/Investigator# 79201, Coburg
  - Site Reference ID/Investigator# 78993, Greenslopes
- Israel (2):
  - Site Reference ID/Investigator# 77860, Afula
  - Site Reference ID/Investigator# 77637, Rehovot
- Site Reference ID/Investigator# 77413, Gdansk, Poland
- Ukraine (5):
  - Site Reference ID/Investigator# 79203, Ivano-Frankivsk
  - Site Reference ID/Investigator# 79205, Khmelnitsky
  - Site Reference ID/Investigator# 79202, Kyiv
  - Site Reference ID/Investigator# 79204, Lviv
  - Site Reference ID/Investigator# 79206, Poltava